CLINICAL TRIAL: NCT05427292
Title: Feasibilty of Serratus Anterior and Pectoral Nerve Blocks (PECS II) Combination as Main Anesthetic Method in Breast Cancer Surgery Patients
Brief Title: Combination of Serratus Anterior and Pectoral Nerve Blocks (PECS II) as Main Anesthetic Method in Breast Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Gamze Ertas, Principal Investigator, Samsun University
Other Study IDs: SamsunU
Record Dates: First submitted 2022-06-13; First posted 2022-06-22 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia
Keywords: regional anesthesia; interfascial plane block; Main anesthetic method

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: serratus anterior block and PECs II block combination — The pre-surgery block will be applied. Sensorial block will be evaluated at the surgical incision site with the pinpirick test at 30 minutes after the block, and if the block is successful, surgery will begin.

SUMMARY:
Aim of this study is to determine the success of combined serratus anterior and PECS-2 block as the main anesthetic method in breast cancer surgery and also to investigate the patient acceptability of this combination and its relationship with surgeon satisfaction.

DETAILED DESCRIPTION:
Breast conserving surgery or mastectomy is applied in the surgical treatment of breast cancer. Axillary interventions range from sentinal lymph node biopsy to lymph node dissection. Clinically significant acute pain develops following breast surgery in 35% of patients.

Today, regional anesthesia is widely used as an opioid-sparing strategy in the treatment of acute postoperative pain. New fascial plane blocks have been developed as alternative or complementary techniques for chest wall analgesia, including pectoral nerve blocks (PECS1-2) and serratus plane block.

In order to reduce the risk of perioperative morbidity and mortality and to meet the patient demand, the demand for awake surgery is increasing in institutions.

Therefore, a prospective observational case series was conducted to explain the efficacy, patient acceptability, and surgeon satisfaction of combined serratus anterior and PECS-2 block as the main anesthetic method for breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-80 and ASA I-III who will undergo unilateral breast cancer surgery will be included in the study.

Exclusion Criteria:

* Patients with previous breast surgery other than excisional biopsy,
* coagulopathy,
* bleeding disease,
* local infection at the injection site,
* history of local anesthetic allergy,
* psychiatric disease (depression, mania, schizophrenia or antipsychotic drug use),
* history of opioid use for more than 4 weeks
* Patients with body mass index (BMI) >40kg/m2 and
* chest deformity (pectus excavatum and pectus carinatum) will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged 18-80 years with breast cancer
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Sufficient surgical anesthesia | up to 30 minutes
  After confirming the sensory block in the surgical area with the post-procedure pinpirick test, successful completion of the surgical procedure 'without the need for deep sedoanalgesia' will be considered 'sufficient surgical anesthesia'.

SECONDARY OUTCOMES:
Pain scores on the Numeric Rating Scale (NRS) | up to 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Quality of recovery 15 scale | up to 24 hours
  Postoperative Quality of Recovery 15 in Turkish scale
analgesic consumption | up to 24 hours
  In the postoperative period, patients will be given opioids according to their pain density with a patient-controlled device, and the daily Morphine consumption in Patient Controlled Analgesia device will be collected
modified Wilson Sedation Scale | up to 2 hours
  1. Oriente, eyes may be closed, but says his name, answers where he is
  2. Sleepy, eyes may be closed, can be warned when called by name
  3. Can be stimulated by mild physical stimulation (earlobe)
  4. Cannot be stimulated by mild physical stimulation
quality of anesthesia | up to 2 hours
  Are you satisfied with the anesthesia? Would you like to have surgery with the same technique again? Would you recommend it to others?
  1. Extremely satisfied,
  2. Satisfied,
  3. Neither satisfied nor dissatisfied,
  4. Not satisfied,
  5. It will be calculated by responding as highly dissatisfied.
scaling working conditions | up to 2 hours
  Working conditions scaling
  Indistinguishable from general anesthesia A little challenging/enough It will be determined by choosing one of the overly challenging/inadequate options.

CONTACTS AND LOCATIONS:
Overall Officials: gamze MD ertaş, specialist, Principal Investigator — Samsun University
Locations (2):
- Turkey (Türkiye) (2):
  - Samsun University, Samsun, Ilkadım
  - Samsun University, Samsun

REFERENCES:
- [Result] Pawa A, Wight J, Onwochei DN, Vargulescu R, Reed I, Chrisman L, Pushpanathan E, Kothari A, El-Boghdadly K. Combined thoracic paravertebral and pectoral nerve blocks for breast surgery under sedation: a prospective observational case series. Anaesthesia. 2018 Apr;73(4):438-443. doi: 10.1111/anae.14213. Epub 2018 Jan 12. PMID 29327341
- [Result] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099